CLINICAL TRIAL: NCT00705692
Title: Effect of Levamisole Supplementation on Tetanus Vaccination Response Rates in Hemodialysis Patients: A Randomized Double-Blind Placebo-Controlled Trial
Brief Title: Effect of Levamisole Supplementation on Tetanus Vaccination Response Rates in Hemodialysis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mohammad mahdi Sagheb, Associate Professor of Medicine, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 86_3893
Record Dates: First submitted 2008-06-24; First posted 2008-06-26 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2013-07

CONDITIONS: Renal Dialysis
Keywords: Tetanus; Vaccines; Renal Dialysis; Levamisole
MeSH Terms: conditions — Tetanus | interventions — Levamisole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levamisole (Experimental): Two 50 mg levamisole tablets daily, six days before and six days after Td vaccination.
  Interventions: Drug: Levamisole
- Placebo (Placebo Comparator): Two placebo tablets daily, six days before and six days after Td vaccination.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levamisole
  Arms: Levamisole
Drug: Placebo
  Arms: Placebo

SUMMARY:
Levamisole as an immunomodulator drug has been demonstrated to improve the immune response to Hepatitis B virus (HBV) vaccination in hemodialysis patients. The aim of this study was to evaluate the effect of levamisole supplementation on tetanus-diphtheria (Td) vaccine response rate in hemodialysis patients.

DETAILED DESCRIPTION:
Levamisole as an immunomodulator drug has been demonstrated to improve the immune response to HBV vaccination in hemodialysis patients. The aim of this study was to evaluate the effect of levamisole supplementation on Td vaccine response rate in hemodialysis patients. In this randomized double-blind placebo-controlled trial 40 hemodialysis patients who had not received tetanus vaccination in a year before investigation and had unprotective anti-tetanus immunoglobulin G (IgG) levels (<0.1 International Unit [IU]/ml) were enrolled. These patients were randomized into two equal groups to receive one dose of intramuscular Td vaccine supplemented with either levamisole 100 mg or placebo daily, six days before and six days after vaccination. The anti-tetanus IgG levels were measured 1 and 6 months after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* being under regular hemodialysis for more than 3 months
* unprotective baseline levels of antitetanus IgG

Exclusion Criteria:

* tetanus diphtheria (Td) vaccination in past year
* leukopenia (WBC<1500 cells/mcL)
* immunosuppressive drug exposure in past 2 months
* recent hospitalization or history of transfusion of blood products in the past 3 months.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-03; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
tetanus seroconversion rate | 1 month and 6 month post vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Mahdi Sagheb, MD, Principal Investigator — Shiaz University of Medical Sciences
Locations (1):
- Faghihi Hospital Hemodialysis Center, Shiraz University of Medical Sciences, Shiraz, Fars, Iran

REFERENCES:
- [Derived] Fallahzadeh MK, Sajjadi S, Singh N, Khajeh M, Sagheb MM. Effect of levamisole supplementation on tetanus vaccination response rates in haemodialysis patients: a randomized double-blind placebo-controlled trial. Nephrology (Carlton). 2014 Jan;19(1):27-31. doi: 10.1111/nep.12158. PMID 24341659